CLINICAL TRIAL: NCT03655379
Title: A Novel Technique for Prediction of Preterm Birth: Fetal Breathing Patterns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University Ankara Hospital (Other)
Collaborators: Batman Maternity Hospital (Unknown)
Responsible Party: Principal Investigator, Sertac Esin, Associate Professor, Baskent University Ankara Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BaskentUAH
Record Dates: First submitted 2018-08-30; First posted 2018-08-31 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Preterm Birth
Keywords: Preterm birth; Fetal nasal Doppler; Fetal breathing
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nasal Doppler (Experimental): Pregnant patients who present with preterm labor will be evaluated with ultrasonography and fetal nasal Doppler will be used to detect specific fetal breathing patterns
  Interventions: Device: Fetal nasal Doppler by ultrasonography

INTERVENTIONS:
Device: Fetal nasal Doppler by ultrasonography — Pregnant patients who present with preterm labor will be evaluated with ultrasonography and fetal nasal Doppler will be used to detect specific fetal breathing patterns and measurements will be performed

SUMMARY:
Preterm birth refers to a delivery that occurs before 37 weeks of gestation. Identification of those who will eventually deliver in the preterm period is very important. However, few interventions have been proven to prolong pregnancy in women at risk such as cervicovaginal fetal fibronectin (fFN) level or transvaginal cervical length measurements. In a meta-analysis comparing fetal breathing with cervicovaginal fetal fibronectin (fFN) level or transvaginal cervical length measurements, absence of fetal breathing was superior to other methods for prediction of preterm birth in 48 hours or 7 days. In this study, the investigators hypothesized that if a fetus holds its breath in case of preterm birth, then there may be specific fetal breathing patterns during preterm labor, which may be detected by ultrasonography

DETAILED DESCRIPTION:
Preterm birth refers to a delivery that occurs before 37 weeks of gestation and it is the leading cause of neonatal morbidity and mortality. 33% of prenatal hospital admissions are due to preterm labor but almost 50% of patients receiving tocolytics in order to prevent birth deliver in the term period. Therefore, identification of those who will eventually deliver in the preterm period is very important. Ideally, identification of modifiable and nonmodifiable risk factors for preterm birth in will lead to interventions that help prevent this complication. However, few interventions have been proven to prolong pregnancy in women at risk such as cervicovaginal fetal fibronectin (fFN) level or transvaginal cervical length measurements. Another method for preterm birth prediction is presence of fetal breathing. In a meta-analysis comparing fetal breathing with cervicovaginal fetal fibronectin (fFN) level or transvaginal cervical length measurements, absence of fetal breathing was superior to other methods for prediction of preterm birth in 48 hours or 7 days. In this study, the investigators hypothesized that if a fetus holds its breath in case of preterm birth, then there may be specific fetal breathing patterns during preterm labor, which may be detected by ultrasonography

ELIGIBILITY:
Inclusion Criteria:

* Pregnant patients between 24-37 gestational weeks with preterm labor : Uterine contractions ≥4 in number in 20 minutes or ≥ 8 in number in 60 minutes and one of the following:
* Cervical dilation ≥ 3 cm
* Transvaginal cervical length <20mm

Exclusion Criteria:

* Multifetal pregnancy
* Cervical dilation > 5 cm
* Heavy vaginal bleeding
* Non-reassuring fetal non-stress test
* Preterm premature rupture of membranes
* Intrauterine growth restriction
* Oligohydramniosis
* Fetal anomaly
* Patients who received tocolytics for preterm labor or corticosteroids for lung maturation
* Drug or substance use which may depress fetal breathing

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Inspiration Duration | Admission ultrasonography
  Fetal Inspiration Duration
Expiration Duration | Admission ultrasonography
  Fetal Expiration Duration

CONTACTS AND LOCATIONS:
Overall Officials: Sertac Esin, M.D., Principal Investigator — Baskent University Medical Faculty; Erhan Okuyan, M.D., Principal Investigator — Batman Kadin Dogum ve Cocuk Hastaliklari Hastanesi
Locations (1):
- Baskent University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Boots AB, Sanchez-Ramos L, Bowers DM, Kaunitz AM, Zamora J, Schlattmann P. The short-term prediction of preterm birth: a systematic review and diagnostic metaanalysis. Am J Obstet Gynecol. 2014 Jan;210(1):54.e1-54.e10. doi: 10.1016/j.ajog.2013.09.004. Epub 2013 Sep 7. PMID 24021995